CLINICAL TRIAL: NCT02342288
Title: Intraoperative Ocular Pressure in Lumbar Spine Fusion Patients
Acronym: IOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Sanford E Emery, MD, MBA, Professor and Chairman WVU Department of Orthopaedics, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 1409441146
Record Dates: First submitted 2015-01-08; First posted 2015-01-19 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-01

CONDITIONS: Raised Ocular Pressure
Keywords: Intraoperative ocular pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Head raised 10 degrees (Experimental): Head raised 10 degrees from neutral position using Gardner Wells tongs
  Interventions: Procedure: Head raised 10 degrees
- Head in neutral position (Active Comparator): Head in neutral position
  Interventions: Procedure: Head in neutral position

INTERVENTIONS:
Procedure: Head raised 10 degrees — Baseline measurement in seated position; anesthetization in the supine position. Prior to turning into the prone position, another measurement was taken. Five minutes after turning prone, a third IOP measurement was obtained. Head was raised to 10 degrees. After 5 minutes a fourth IOP measurement was performed. Repeat measurements were taken every 15 minutes until three sequential measurements were within plus or minus 3 mmHg of one another; thereafter, measurements were obtained every hour until end of case. A final measurement was taken after turning the patient supine and 5 minutes elapsed for equilibration.
  Arms: Head raised 10 degrees
Procedure: Head in neutral position — Baseline measurement in seated position; anesthetization in the supine position. Prior to turning into the prone position, another measurement was taken. Five minutes after turning prone, a third IOP measurement was obtained. After 5 minutes a fourth IOP measurement was performed. Repeat measurements were taken every 15 minutes until three sequential measurements were within plus or minus 3 mmHg of one another; thereafter, measurements were obtained every hour until end of case. A final measurement was taken after turning the patient supine and 5 minutes elapsed for equilibration.
  Arms: Head in neutral position

SUMMARY:
A rare but terrible complication of vision loss has been known to occur after surgery, including spine surgery. It is commonly thought that increased intraocular pressure (IOP) is one of the reasons for this rare vision loss. It has been shown that the prone position can increase the IOP, and that tilting the patient with the head down can also increase IOP. The investigators will be measuring IOP before, during, and after a posterior spine surgery to see if the investigators can influence the intraocular pressure with elevated head position change. Two groups will be studied: one group of patients will receive standard care with the head in neutral position, while the other group will have the head slightly elevated 10 degrees during prone spine surgery.

DETAILED DESCRIPTION:
It has been reported that postoperative vision loss after lumbar surgery is increasing. It is an uncommon but devastating complication. One of the risk factors that has been reported is increased intraocular pressure (IOP), which may decrease perfusion pressure to the optic nerve. Intraocular pressure in anesthetized, prone spine patients has been studied with the head in neutral position. The prone position and duration of the procedure did increase the IOP. Our hypothesis is that adjusting the position of the head in space will alter the intraocular pressure, with an extended position decreasing IOP. This study is a, randomized, controlled design: neutral head position (standard care) or extended head position (intervention group). Patients who qualify for spinal fusion surgery and meet the inclusion criteria will be randomized to either the neutral (standard practice) or the intervention group.Randomization of patients will be computer generated.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective lumbar spinal fusion surgery; ages 18-80

Exclusion Criteria:

* Less than 18 years of age
* Glaucoma, previous eye surgery, eye injury, or eye trauma, cervical myelopathy, prior cervical spine surgery, current neoplasm, patients who have neck pain with 10 degrees active extension.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2008-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanford E Emery, MD, MBA, Principal Investigator — West Virginia University

IPD SHARING:
Plan to Share IPD: No
Group data will be published. Not individual data.

REFERENCES:
- [Background] Ozcan MS, Praetel C, Bhatti MT, Gravenstein N, Mahla ME, Seubert CN. The effect of body inclination during prone positioning on intraocular pressure in awake volunteers: a comparison of two operating tables. Anesth Analg. 2004 Oct;99(4):1152-1158. doi: 10.1213/01.ANE.0000130851.37039.50. PMID 15385367
- [Background] Carey TW, Shaw KA, Weber ML, DeVine JG. Effect of the degree of reverse Trendelenburg position on intraocular pressure during prone spine surgery: a randomized controlled trial. Spine J. 2014 Sep 1;14(9):2118-26. doi: 10.1016/j.spinee.2013.12.025. Epub 2014 Jan 20. PMID 24456677
- [Background] Walick KS, Kragh JE Jr, Ward JA, Crawford JJ. Changes in intraocular pressure due to surgical positioning: studying potential risk for postoperative vision loss. Spine (Phila Pa 1976). 2007 Nov 1;32(23):2591-5. doi: 10.1097/BRS.0b013e318158cc23. PMID 17978659
- [Derived] Emery SE, Daffner SD, France JC, Ellison M, Grose BW, Hobbs GR, Clovis NB. Effect of Head Position on Intraocular Pressure During Lumbar Spine Fusion: A Randomized, Prospective Study. J Bone Joint Surg Am. 2015 Nov 18;97(22):1817-23. doi: 10.2106/JBJS.O.00091. PMID 26582611

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in the orthopaedic clinic at West Virginia University beginning November 2008 and recruitment ended February 2014.
Pre-assignment Details: Seventy-nine patients were consented and enrolled. Sixty-three were randomized. Twenty-seven patients did not complete the study. Of the 27, 16 were never randomized. The number of patients who were randomized, started the study and received full treatment or placebo was 52.
  Reasons are listed below for those who did not complete the study.
Period: Overall Study
Arm/Group | Head Raised 10 Degrees | Head in Neutral Position
Started | 30 (16 patients were not randomized to either arm.) | 33 (various issues listed below caused removal of subjects)
Completed | 25 | 27
Not Completed | 5 | 6
Not completed — no protocol anesthesiologist available | 3 | 2
Not completed — anesthesia leak in system | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — coordinator contaminated with blood | 0 | 1
Not completed — subject cannot tolerate numbing drops | 0 | 1
Not completed — coordinator not available | 0 | 2

BASELINE CHARACTERISTICS:
Population: no significant differences in baseline demographics between the groups
Groups:
- Total: Total of all reporting groups
Arm/Group | Head Raised 10 Degrees | Head in Neutral Position | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 17 | 37
  >=65 years | 5 | 10 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 8 | 9 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 25 | 27 | 52
Region of Enrollment [Number; unit: participants]
  United States | 25 | 27 | 52

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraoperative Ocular Pressure in Lumbar Spine Fusion Patients Head Raised 10 Degrees or Kept in Neutral Position
Description: The objective is to determine if slight elevation of the head (10 degrees up from neutral) can decrease the IOP compared to remaining in neutral position (standard of care) for the entire surgery. The mean values for Δ IOP measurements (i.e. two eye average maximum IOP - two eye average baseline IOP obtained at first prone measurement).
Time Frame: Prone; 5 minutes after head raised to 10 degrees; every 15 minutes; 1 hr until end of surgery
Population: Subjects who were undergoing elective lumbar spine surgery.
Measure: Mean (95% Confidence Interval); unit: mm Hg
Groups:
- Head Raised 10 Degrees: Head raised 10 degrees from neutral position using Gardner Wells tongs
  Head raised 10 degrees: Five minutes after turning prone, an IOP measurement was obtained. Head was raised to 10 degrees. After 5 minutes an IOP measurement was performed. Repeat measurements were taken every 15 minutes until three sequential measurements were within plus or minus 3 mmHg of one another; thereafter, measurements were obtained every hour until end of case. A final measurement was taken after turning the patient supine and 5 minutes elapsed for equilibration.
- Head in Neutral Position: Head in neutral position
  Head in neutral position: Five minutes after turning prone, an IOP measurement was obtained. After 5 minutes an IOP measurement was taken. Repeat measurements were taken every 15 minutes until three sequential measurements were within plus or minus 3 mmHg of one another; thereafter, measurements were obtained every hour until end of case. A final measurement was taken after turning the patient supine and 5 minutes elapsed for equilibration.
Arm/Group | Head Raised 10 Degrees | Head in Neutral Position
Number analyzed (Participants) | 25 | 27
mm Hg | 9.26 [6.65 to 11.87] | 13.79 [10.60 to 16.97]

2. Secondary Outcome: Change and Correlations in Intraoperative Ocular Pressure in Lumbar Spine Fusion Patients
Description: The secondary outcome is to evaluate factors (age, gender, duration of procedure, blood loss, intraoperative fluids, blood pressure, and carbon dioxide levels) looking for correlations with intraocular pressure changes.
Time Frame: prone; every 15 minutes; 1 hr until end of surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: One year
Description: Follow up occurred at 2 weeks, 1 month, 3 month, 6 months, and 1 year.
Arm/Group | Head Raised 10 Degrees | Head in Neutral Position
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 1/25 | 0/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Head Raised 10 Degrees (N=25) | Head in Neutral Position (N=27)
mild corneal abrasion (Eye disorders) | 1 (1) | 0 (0) — One patient sustained a mild corneal abrasion that resolved in 24 hours using ophthalmic ointment.

LIMITATIONS AND CAVEATS:
The main limitation of our trial is that these were not consecutive cases, due to availability of the technician and a limited number of anesthesiologists on the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No